CLINICAL TRIAL: NCT01893047
Title: Effect of Quiet or Listening to Music While Breastfeeding on the Production and Lipid and Sodium Content of the Milk
Brief Title: Effect of Music on Breastmilk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Professor, Department of Pediatrics, Neonatology, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 47585; University of Rochester (Other: University of Rochester)
Record Dates: First submitted 2013-06-20; First posted 2013-07-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Milk Production
Keywords: breast milk production

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- no music (No Intervention): The mother will be randomized to receive each od three experimental conditions: live music, recorded music, no music in random order over the course of three pumping sessions. She will then experience all three conditions again in random order
- live music (Experimental): The mother will be randomized to receive each od three experimental conditions: live music, recorded music, no music in random order over the course of three pumping sessions. She will then experience all three conditions again in random order
  Interventions: Behavioral: live music
- recorded music (Experimental): The mother will be randomized to receive each od three experimental conditions: live music, recorded music, no music in random order over the course of three pumping sessions. She will then experience all three conditions again in random order
  Interventions: Behavioral: recorded music

INTERVENTIONS:
Behavioral: live music — live harp music
  Arms: live music
Behavioral: recorded music — recorded harp music
  Arms: recorded music

SUMMARY:
A mother of a preterm infant listening to music while pumping her breasts will produce more milk than a similar mother who is not listening to music. A mother listening to live music will produce more milk than a mother listening to recorded music

DETAILED DESCRIPTION:
1. Purpose of the study. The purpose of this study is to determine whether listening to music under three conditions: (1) when a music practitioner is playing background harp music, (2) when a CD is playing exactly the same background harp music, or (3) when no background music is being played will have an effect on the flow, lipid (fat), or the sodium content of breast milk.

PRIMARY HYPOTHESES: (1) A primiparous mother of a preterm infant listening to music while pumping her breasts will produce more milk than a similar mother who is not listening to music. (2) A mother listening to live music will produce more milk than a mother listening to recorded music.

EXPLORATORY HYPOTHESIS: (1) The milk of a mother listening to music while pumping her breasts will have higher lipid content and lower sodium content than a mother who is not listening to music.

PRIMARY OBJECTIVE: This pilot study will investigate the feasibility of measuring the amount of breast milk produced by mothers who are pumping breast milk for their preterm infant under one of three conditions: (1) when a music practitioner is playing background harp music, (2) when a CD is playing exactly the same background harp music, or (3) when no background music is being played.

II. CHARACTERISTICS OF THE RESEARCH POPULATION

1. Number of Subjects. There will be a total number of 40 mothers participating in this study.
2. Gender of Subjects. All subjects will be female. Men cannot express breast milk.
3. Age of Subjects. Mothers will be between the ages of 18 and 45. Mothers under the age of 18 are excluded because they are minors. Ages 18 to 45 are the typical ages that women give birth.
4. Racial and Ethnic Origin. The racial and ethnic distribution of the subjects are expected to reflect the general population of mothers between the ages of 18 and 45 who deliver preterm infants at Strong Memorial Hospital.
5. Inclusion Criteria. First time mothers between the ages of 18 and 45 who have had a vaginal or caesarean delivery and are feeling well. First time mothers are used to avoid confounding variables due to previous positive or negative experiences from expressing milk. Their infant will have been born at less than 32.0 weeks of gestation. Mothers will intend to breastfeed and are planning to pump milk on site in the NICU at least once/day and will be recruited 7-10 days postpartum. Mothers who smoke, are taking medication that may interfere with breastfeeding, and who have undergone prior breast surgery will not be excluded since they are their own control. With regard to language, mothers must be able to understand the directions and sign a consent form in English.
6. Exclusion Criteria. Mothers will not be recruited whose infant has a low likelihood of survival as determined by the attending physician. Mothers who have been diagnosed with mastitis will not be recruited for the study.
7. Vulnerable Subjects. No vulnerable subjects will be included in this study.

III. METHODS AND PROCEDURES

1. Methods and Procedures. : After a mother has agreed to participate, she will complete the informed consent process and then complete the baseline questionnaire (pre-session 1).

   Only one breast pumping session will be assessed on a given day. All remaining breast pumping sessions on any given day conducted by the mother per her daily routine will not be a part of the study and no data will be collected at those times.

   Study Session 1 (Orientation): The mother will arrive at the pumping room and get comfortably settled. The mother will be asked to turn off all electronic equipment (cell phone, iPod). Reading material such as Good Housekeeping, Better Homes and Gardens, and Parents magazines will be available for her use if she wishes. She will attach one or both breasts to the Symphony Breast pump by Medela that is in standard usage in the NICU. (Note: Mother will decide if she will pump one or both breasts at a time. Whatever condition she chooses will remain the same throughout all study sessions.) Recorded music will be played for this session. While the breast pump is being applied, a third female person will enter the room and remain behind a privacy screen. This third person will either be a research assistant, physician, or nurse who will be trained in patient confidentiality and the rights of research subjects. When the breast pump is applied, the third person will start the recorded music. She will have no communication with the mother or the research assistant.

   The mother will then pump her breast(s) into an 80 cc volufeed container. The research assistant will sit behind the mother facing away from the mother while the mother is pumping and will time the pumping for 15 minutes. The amount of milk produced during the 15 minute period will be measured and recorded by the research assistant. To ensure that the mother can meet her baby's needs, a 2 cc aliquot will only be taken if 10 cc has been produced in 15 minutes; and if including the current pumping session, there is sufficient milk for 24 hours of infant feeding. If the previous two conditions are met, a lactation consultant or the mother's nurse will remove a 2 cc aliquot at the end of the session. The 2 cc aliquot will be frozen for future analysis. If the previous two conditions are not met, a 2 cc aliquot will not be taken and this will be noted on the data collection sheet. The remaining milk will be combined with any additional milk the mother may produce during the remainder of the pumping session. She will label and store the milk for later use by her infant according to her usual routine. When the mother tells the research assistant that she has completed pumping, the third person will quietly leave the room.

   The mother will then be randomized to receive each of the three experimental conditions (live music, recorded music, and no music) in random order over the course of three pumping sessions. She will then experience all three conditions again in random order (a three-block pattern randomized twice.) Study Sessions 2-7: The mother will arrive at the pumping room and become comfortably settled. The mother will be asked to turn off all electronic equipment (cell phone, iPod). Reading material such as Good Housekeeping, Better Homes and Gardens, and Parents magazines will be available for her use if she wishes. She will attach one or both breasts to the Symphony Breast pump by Medela that is in standard use in the NICU. (Note: Mother will decide if she will pump one or both breasts at a time. Whatever condition she chooses will remain the same throughout all study sessions.) The mother will not be told whether live, recorded, or no music is played during her session. While the breast pump is being applied, a third female person will enter the room and remain behind a privacy screen. If live music is played, this third person will be the musician. In order to provide the same conditions even when music is not played, a third female will still enter the room and remain behind the privacy screen. She will have no communication with the mother or the research assistant.

   At that point, either live music, recorded music, or no music will be played. When music is played, the same music will be played at each session. The mother will pump her breast(s) into an 80 cc volufeed container. The research assistant will sit behind the mother facing away from the mother while the mother is pumping and will time the pumping for 15 minutes. The amount of milk produced during the 15-minute period will be measured and recorded by the research assistant on a data collection sheet. To ensure that the mother can meet her baby's needs, a 2 cc aliquot will be taken only if 10 cc has been produced in 15 minutes; and if including the current pumping session, there is sufficient milk for 24 hours of infant feeding . If the previous two conditions are met, a lactation consultant or the mother's nurse will remove a 2 cc aliquot at the end of the session. The 2 cc aliquot will be frozen for future analysis. If the previous two conditions are not met, a 2cc aliquot will not be taken and this will be noted on the data collection sheet. The remaining milk will be combined with any additional milk the mother may produce during the remainder of the pumping session. She will label and store the milk for later use by her infant according to her usual routine. When the mother tells the research assistant that she has completed pumping, the third person will stop playing, turn off the player, and/or simply quietly leave the room.

   ASSESSMENTS (attached): Mothers will complete a Pre-session 1 (orientation) questionnaire that will provide general demographic information as well as information about mother's reasons for and plans for the duration of breastfeeding. The research assistant will complete a questionnaire with the mother's assistance as appropriate after each subsequent session (2-7). Assessments session 2-7 inquire about the session as well as the mother's emotional state. The mother will complete a final questionnaire after session 7 regarding her experiences with live music, recorded music, and quiet while pumping her breasts. The fat content and sodium content of all breast milk samples obtained during sessions 2-7 will be measured.
2. Data Analysis and Monitoring. The mother will serve as her own control. Milk produced over 15 minutes will be measured during each session and the amount of milk produced during the two sessions under identical conditions will be averaged. The primary outcome will be the differences in the amount of milk produced by the mother under each of the three conditions.

   We will use 40 subjects, with each subject being her own control. This sample size will allow us to detect an effect size of 0.5, assuming a paired t-test and a Bonferroni-corrected p value of 0.025 (to account for two primary comparisons). We will use factorial repeated measures ANOVA - "condition" (live music, recorded music, no music) as the main effect to be examined. We will run contrasts to examine the two hypotheses. Since each mother will act as her own control, we will be examining within-subject differences. Thus, infant age, weight, and medical condition will be internally controlled and will not be included in the analyses. However, variables such as the mother's emotional and physical condition and time since last pumping, which could change day-to-day, could be included in our modeling, if there is significant within-subject variance.

   The sodium content of the milk will be measured using standard clinical laboratory procedures. Lipid (fat) content of milk will be measured using the creamatocrit (10).
3. Data Storage and Confidentiality. Data will be entered into a password-protected encrypted electronic database accessible only to study personnel. All print/paper forms will be kept in a locked filed in a locked office in a limited accessibility suite.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers between the ages of 18 and 45 who have had a vaginal or caesarean delivery and are feeling well.
* First time mothers are used to avoid confounding variables due to previous positive or negative experiences from expressing milk. Their infant will have been born at less than 32.0 weeks of gestation.
* Mothers will intend to breastfeed and are planning to pump milk on site in the NICU at least once/day and will be recruited 7-10 days postpartum.
* Mothers who smoke, are taking medication that may interfere with breastfeeding, and who have undergone prior breast surgery will not be excluded since they are their own control.
* With regard to language, mothers must be able to understand the directions and sign a consent form in English.

Exclusion Criteria:

* Mothers will not be recruited whose infant has a low likelihood of survival as determined by the attending physician.
* Mothers who have been diagnosed with mastitis will not be recruited for the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Volume of milk in ten minutes | 10 days
  Milk volume in Ml.

SECONDARY OUTCOMES:
Milk sodium | 10 days
  Sodium in Meq/L.
Milk lipid | 10 days
  Milk triglycerides and cholesterol in Mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lawrence, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States